CLINICAL TRIAL: NCT07184255
Title: Multilingual Animated Video Education for Retinal Detachment Surgery: A Randomized Controlled Trial
Brief Title: Animated Video Education for Retinal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Tina Felfeli, Doctor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-5893
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Retinal Detachment
Keywords: Retinal Detachment; Patient Education; Multilingual Video Intervention; Health Literacy; Eye surgery; Knowledge translation
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, 1:1 randomization, stratified by surgical procedure (PnR, PPV, SB) and language proficiency (English vs non-English).
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Standard Counselling) (No Intervention): Standard pre-operative verbal counselling by ophthalmologist/clinic staff.
- Intervention Arm (Video + Standard Counselling) (Experimental): Standard counselling plus a 5-minute animated video in the patient's preferred language, covering diagnosis, surgical steps, and post-operative positioning. Video includes high-contrast visuals and audio narration.
  Interventions: Other: Patient Education Video Intervention

INTERVENTIONS:
Other: Patient Education Video Intervention — Animated video with high-contrast visuals and audio narration in the patient's preferred language, covering diagnosis, surgical steps, and post-operative positioning.
  Arms: Intervention Arm (Video + Standard Counselling)

SUMMARY:
Retinal detachment is a vision-threatening condition that requires urgent surgical repair. Understanding the condition, the surgery, and post-operative instructions is difficult for many patients, particularly in multilingual and multicultural populations. This study will evaluate whether short, animated educational videos, available in 25 languages and designed with accessibility features for patients with low vision, improve patient knowledge, reduce anxiety, and support adherence to post-operative instructions when added to standard counselling. Patients will be randomized to standard counselling alone versus counselling plus video in their preferred language. Outcomes will be measured with validated questionnaires at baseline, immediately after counselling, and one week post-surgery.

DETAILED DESCRIPTION:
Retinal detachment is a surgical emergency that can result in irreversible vision loss if untreated. Surgical options include pneumatic retinopexy, pars plana vitrectomy, and scleral buckle. Successful outcomes depend not only on timely surgery but also on patient understanding of their condition, the procedure, and critical post-operative instructions, especially positioning requirements. Traditional verbal counselling can be difficult for patients to absorb, particularly in multicultural populations where language barriers and variable health literacy are common.

This trial will evaluate a multilingual, animated educational video intervention designed to address these challenges. Each video is five minutes in length and includes simplified explanations of retinal detachment, key surgical steps, and post-operative positioning. Accessibility features such as high-contrast visuals, bold graphics, and audio narration allow use by patients with varying levels of vision and literacy. The videos are available in 25 languages, selected to reflect the most commonly spoken languages in Canada and globally.

Participants will be randomized to receive either standard counselling alone or counselling plus video in their preferred language. Outcomes include knowledge acquisition, anxiety reduction, and adherence to positioning instructions, measured with validated questionnaires. Findings will inform scalable strategies to improve patient education, promote equity in ophthalmic care, and reduce preventable complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Diagnosis of primary rhegmatogenous retinal detachment.
* Planned repair with pneumatic retinopexy (PnR), pars plana vitrectomy (PPV), or scleral buckle (SB).
* Able to provide informed consent.
* Preferred language available among study videos.

Exclusion Criteria:

* Repeat retinal detachment surgery in study eye.
* Combined complex procedures (e.g., PPV + corneal transplant).
* Severe cognitive impairment precluding consent.
* Hearing impairment preventing use of audio track (without aid).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 1 week
  Change in knowledge score (0-10 scale) from baseline (pre-surgery) to post-intervention and procedure.

SECONDARY OUTCOMES:
Anxiety | 1 week
  Change in anxiety score (0-10 visual analog scale) from baseline to post-intervention and 1 week post-surgery.
Understanding | 1 week
  Change in self-reported understanding and self-efficacy (0-10 scale).
Adherence | 1 week
  Adherence to post-operative positioning (self-reported hours/day, categorical scale) at 1 week.
Patient Satisfaction | 1 week
  Patient satisfaction with information received (Likert 5-point scale) at 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Yes. De-identified individual-level data (survey responses, knowledge scores, anxiety scales) will be shared via institutional repositories upon reasonable request, following UHN REB approval.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months of publication.